CLINICAL TRIAL: NCT03163355
Title: Comparison of Pureed Rice Using a Gelling Agent and Standard Pureed Rice in Swallowing in Elderly Patients With Dysphagia
Brief Title: Comparison of Pureed Rice Using a Gelling Agent and Standard Pureed Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017VE
Record Dates: First submitted 2017-05-20; First posted 2017-05-23 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Swallowing Disorder
Keywords: pureed diet; dysphasia
MeSH Terms: conditions — Deglutition Disorders; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pureed rice with a gelling agent (Active Comparator): 3 ml of pureed rice containing a gelling agent is attempted to swallow under endoscopic examination of swallowing
  Interventions: Other: a gelling agent
- standard pureed rice (Placebo Comparator): 3 ml of standard pureed rice is attempted to swallow under endoscopic examination of swallowing
  Interventions: Other: a gelling agent

INTERVENTIONS:
Other: a gelling agent — Pureed rice containing a gelling agent (Softia U, Nutri Co., Ltd., Yokkaichi, Japan) is compared with the standard purred rice in the condition of swallowing.

SUMMARY:
The texture of the pureed diet is likely to be most useful factor predictive of the prevention of aspiration pneumonia. However, it has not been previously reported what kinds of texture of the pureed diet can prevent aspiration pneumonia. Using endoscopic swallowing evaluation, we attempt to compare two kinds of the pureed diets to choose the better texture of pureed diets in elderly patients with severe dysphagia.

DETAILED DESCRIPTION:
The degree of dysphagia is evaluated using Hyodo.Komagane score (0-12). Subsequently, a randomized, crossover trial using pureed rice containing a gelling agent (Softia U, Nutri Co., Ltd., Yokkaichi, Japan), or standard pureed rice is performed in patients with dysphagia.

The extent of pharyngeal clearance after swallowing of each pureed rice and test jelly (Isotonic green jelly®, Nutri Co., Ltd., Yokkaichi, Japan) is scored as follows:

1. No remains
2. Pharyngeal clearance is obtained after swallowing of test jelly once
3. Pharyngeal clearance is obtained after swallowing of test jelly twice
4. Pharyngeal clearance is obtained after swallowing of test jelly three times and more
5. In spite of swallowing of test jelly, pharyngeal residues remain and/or penetrate into larynx.

Evaluation Primary outcome: The pharyngeal clearance score (1-5) Secondary outcome: Patient feeling regarding pharyngeal clearance after the swallowing of pureed rice and/or test jelly (0 remains -100% complete clearance)

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients who underwent endoscopic swallowing evaluation at Showa Inan General Hospital

Exclusion Criteria:

* an age less than 65 years old or the presence of an acute infection.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
The pharyngeal clearance score (1-5) | 24 months
  1. No remains
  2. Pharyngeal clearance is obtained after swallowing of test jelly once
  3. Pharyngeal clearance is obtained after swallowing of test jelly twice
  4. Pharyngeal clearance is obtained after swallowing of test jelly three times and more
  5. In spite of swallowing of test jelly, pharyngeal residues remain and/or penetrate into larynx.

SECONDARY OUTCOMES:
Patient feeling regarding pharyngeal clearance | 24 months
  Patient feeling regarding pharyngeal clearance after the swallowing of pureed rice and/or test jelly (0 remains -100% complete clearance)

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No